CLINICAL TRIAL: NCT01315028
Title: A Pilot Randomised Controlled Trial of Cognitive Behaviour Therapy for Early Bipolar Disorder
Brief Title: Bipolar Intervention Study: Cognitive Interpersonal Therapy
Acronym: BISCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government); University of Glasgow (Other)
Responsible Party: Principal Investigator, Jamie Kirk, Clinical Psychologist / Chief Investigator, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN09CP546; CZG/2/472 (Other Grant/Funding Number: Chief Scientist Office, Scottish Executive)
Record Dates: First submitted 2011-03-07; First posted 2011-03-15 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-04

CONDITIONS: Mania; Hypomania; Bipolar Affective Disorder
Keywords: mania; hypomania; bipolar affective disorder; psychological intervention; cognitive therapy
MeSH Terms: conditions — Mania; Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychological Therapy (Experimental): Cognitive Interpersonal Therapy (CIT) was a psychological therapy which emphasised assessment, engagement and formulation; normalizing and compassionate understanding; specific cognitive-behavioural and interpersonal strategies; self-management and social rhythm regulation; affect regulation, and staying well (Gumley & Schwannauer, 2006).
  Interventions: Other: Cognitive Interpersonal Therapy
- Treatment As Usual (Active Comparator): All participants continued to receive their usual care from their local community mental health team and other psychological therapies were not withheld during the conduct of the trial.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: Cognitive Interpersonal Therapy — Cognitive Interpersonal Therapy in Early Bipolar Disorder: Individuals will receive up to six months of individual CIT-BP. CBT will emphasise assessment, engagement and formulation; normalizing and compassionate understanding; specific cognitive and behavioural strategies; self-management and social rhythm regulation; affect regulation, and staying well (Gumley & Schwannauer, 2006).
  Other Names: Psychological Therapy
  Arms: Psychological Therapy
Other: Treatment As Usual — The comparison group is treatment as usual (TAU). This will comprise of the individuals normal psychiatric care and will vary with individual and locality and is therefore not specified.
  Other Names: Normal clinical care
  Arms: Treatment As Usual

SUMMARY:
There is a need to develop a better understanding of the early phase of bipolar disorder, and to develop and evaluate effective psychosocial interventions that assist people in this phase. The purpose of this study is to determine whether or not it is feasible to conduct a larger study of the effectiveness of cognitive interpersonal therapy (a psychological therapy) with individuals who have experienced their first or second treated episode of mania or hypomania (symptoms common in early development of bipolar disorders).

DETAILED DESCRIPTION:
The 'PICO' framework (Oxman, Sackett, and Guyatt, 1993; Richardson, Wilson, Nishikawa, and Hayward; 1995) was used to specify the parameters of the study aims and objectives:

1. Population: could appropriate individuals be identified and recruited to a trial of CIT for early bipolar disorder?
2. Intervention: would CIT be an acceptable intervention for individuals following a first or second treated episode of mania and or hypomania? Could we identify any modifications required to the CIT protocol used with this group?
3. Control group: could an appropriate group of participants be recruited to facilitate a comparison with the CIT intervention? Could we explicitly establish the usual care package and its local implementation?
4. Outcomes: which outcomes are appropriate for measuring relevant dimensions of a treatment effect?

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals will have experienced their first or second treated episode of mania and / or hypomania in the previous 12-months prior to study entry.

Exclusion Criteria:

* Participants will be excluded if there is a (1) diagnosis of learning disability; (2) inability to participate in psychotherapy/research due to acute medical condition or acute mania

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie D Kirk, D.Clin.Psy, Principal Investigator — NHS Greater Glasgow & Clyde / University of Glasgow; Andrew I Gumley, PhD, Study Chair — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Gartnavel Royal Hospital, Glasgow, Lanarkshire
  - NHS Greater Glasgow & Clyde, Glasgow

REFERENCES:
- See also: Study webpage — http://www.gla.ac.uk/departments/mentalhealthandwellbeing/biscit/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consecutively recruited from mental health services within the Glasgow. A total of 32 patients were referred to the study during the 9-month recruitment window between November 2010 and July 2011 (3.5 referrals/month). Of the 32 patients referred 23 consented to participate in the trial. This equates to a consent rate of 71.88%.
Pre-assignment Details: Of the 32 individuals referred, 6 were not assessed as: 3 refused consent, 2 were unable to be contacted within recruitment window and 1 individual moved away from the study location. A further three individuals did not meet our inclusion criteria.
Groups:
- Psychological Therapy: Cognitive Interpersonal Therapy : Cognitive Interpersonal Therapy in Early Bipolar Disorder: Individuals will receive up to six months of individual CIT-BP. CBT will emphasise assessment, engagement and formulation; normalizing and compassionate understanding; specific cognitive and behavioural strategies; self-management and social rhythm regulation; affect regulation, and staying well (Gumley & Schwannauer, 2006).
- Treatment As Usual: Normal Clinical Care : The comparison group is treatment as usual (TAU). This will comprise of the individuals normal psychiatric care and will vary with individual and locality and is therefore not specified.
Period: Overall Study
Arm/Group | Psychological Therapy | Treatment As Usual
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychological Therapy | Treatment As Usual | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.40 (6.90) | 41.60 (45.50) | 37.5 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS) (Montogomery and Asberg, 1979)
Description: The Montgomery Asberg Depression Rating Scale (MADRS) (Montgomery and Asberg, 1979) is a semi-structured interview designed to assess the presence and severity of 10 core symptoms of depression. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  The questionnaire includes questions on the following symptoms 1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts. Usual cutoff points are:
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: Baseline to End of Study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychological Therapy | Treatment As Usual
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 26.20 (12.12) | 20.20 (13.92)
  End of Study | 16.11 (11.82) | 15.22 (16.66)
Statistical Analysis 1: Comparison: Psychological Therapy vs Treatment As Usual; Test type: Superiority or Other; p = 0.05, ANOVA

2. Primary Outcome: Bech-Rafaelsen Mania Rating Scale (BRMS) [Bech et al, 1979]
Description: The Bech-Rafaelsen Mania Rating Scale (BRMS) [Bech et al, 1979] provides a structured format for a clinician to assess the presence and severity of 11 core symptoms of hypomania or mania.Higher BRMS score indicates more severe symptoms of mania, and each item yields a score of 0 to 4. The overall score ranges from 0 to 44. Usual cutoff points are:
  0 to 15 - normal /symptom absent 15 to 20 - mild 21 to 28 - moderate >34 - severe
Time Frame: Baseline to End of Study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychological Therapy | Treatment As Usual
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 6.00 (7.76) | 6.70 (4.42)
  End of Study | 4.78 (4.55) | 4.11 (5.09)
Statistical Analysis 1: Comparison: Psychological Therapy vs Treatment As Usual; Parametric and non-parametric descriptive data were summarised and presented. All data analyses were based on the Intention to Treat (ITT) principle. For the main analysis, Repeated Measures Analysis of Variance was performed to identify signals suggesting treatment effects on the outcome measures. Effect sizes were also calculated in order to further examine suggestive trends in the data indicating appropriate outcomes for further research; Test type: Superiority or Other; p = 0.996, ANOVA

3. Secondary Outcome: The Internal State Scale (ISS) (Bauer et al, 1991)
Description: The Internal State Scale (ISS) (Bauer et al, 1991) is a 15 item self-report scale that utilizes 100 mm visual analogue scales to assess the presence and severity of symptoms, ranging from 'not at all / rarely' to 'very much so / much of the time' (score range per item 0 to 100). The ISS assesses depressive and hypomanic / manic symptoms across four factors: perceived conflict, activation, well-being and depression. Perceived Conflict is assessed across 5 items (score range 0 to 500), Activation across 5 items (score range 0 to 500), Well-being across 3 items (score range 0 to 300) and Depression across 2 items (score range 0 to 200).
  The Well-being subscale is used in conjunction with the Activation subscale for mood state discrimination. The suggested scoring algorithm is as follows:
  Mood State Activation Subscale Score Well-Being Subscale Score (Hypo)Mania >155 >125 Mixed State >155 <125 Euthymia <155 >125 Depression <155
Time Frame: monthly until October 2011
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychological Therapy | Treatment As Usual
Number analyzed (Participants) | 9 | 9
units on a scale
  ISS - Perceived Conflict (Baseline) | 126.00 (94.78) | 78.00 (62.32)
  ISS - Well-being (Baseline) | 97.00 (63.08) | 181.00 (53.84)
  ISS - Activation (Baseline) | 122.00 (81.89) | 114.00 (86.31)
  ISS - Depression (Baseline) | 76.00 (68.02) | 41.00 (50.21)
  ISS - Perceived Conflict (End of Study) | 142.00 (94.84) | 94.44 (105.37)
  ISS - Well-being (End of Study) | 127.78 (67.97) | 137.78 (82.73)
  ISS - Activation (End of Study) | 131.11 (108.45) | 113.33 (117.69)
  ISS - Depression (End of Study) | 46.64 (47.17) | 45.56 (57.69)
Statistical Analysis 1: Comparison: Psychological Therapy vs Treatment As Usual; Test type: Superiority or Other; p < 0.05, ANOVA

4. Secondary Outcome: Global Assessment of Functioning (GAF)
Description: Participant functioning was assessed using the Global Assessment of Functioning (GAF) (APA, 1987). The Global Assessment of Functioning (GAF) is a numeric scale (0 through 100) used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of adults, e.g., how well or adaptively one is meeting various problems-in-living, with higher score indicating higher functioning. The score is often given as a range, from 1 - 10 Persistent danger of severely hurting self or others (e.g., recurrent violence) or persistent inability to maintain minimal personal hygiene or serious suicidal act with clear expectation of death, to 91 - 100 No symptoms. Superior functioning in a wide range of activities, life's problems never seem to get out of hand, is sought out by others because of his or her many positive qualities.
Time Frame: monthly until October 2011
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychological Therapy | Treatment As Usual
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline | 57.90 (20.40) | 60.90 (10.37)
  End of Study | 72.00 (14.05) | 70.56 (16.45)
Statistical Analysis 1: Comparison: Psychological Therapy vs Treatment As Usual; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Psychological Therapy | Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychological Therapy (N=10) | Treatment As Usual (N=10)
Suicide (Psychiatric disorders) | 0 (0) | 1 (1) — One participant randomized to TAU completed suicide
Admission to psychiatric Hospital (Psychiatric disorders) | 0 (0) | 1 (1) — One participant randomized to TAU group was admitted to psychiatric hospital.

LIMITATIONS AND CAVEATS:
A definitive clinical trial should incorporate an appropriate sample size, incorporate more than one therapist, assess fidelity and competence in therapy delivery and also include measurements of health economic dimensions of outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes